CLINICAL TRIAL: NCT00641797
Title: A Randomized Trial to Evaluate Resolution of Symptoms Using Vestibular Rehab Versus Conventional Therapy in Patients Presenting to the Emergency Department (ED) With Diagnosis of Benign Paroxysmal Positional Vertigo (BPPV)
Brief Title: Treating Benign Paroxysmal Positional Vertigo (BPPV) in ED Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, David Burmeister, Chair, Department of Emergency Medicine, Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-2006123IRB#
Record Dates: First submitted 2008-02-13; First posted 2008-03-24 (Estimated); Results first posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Benign Paroxysmal Positional Vertigo
Keywords: Canalith Repositioning Technique; Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo | interventions — Meclizine; Lorazepam; Diazepam; Diphenhydramine; Ondansetron

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1, Conventional Therapy (Active Comparator): Patients will receive standard conventional medication therapy (i.e., meclizine, diphenhydramine, lorazepam, ondansetron).
  Interventions: Drug: Meclizine; Drug: Lorazepam; Drug: Diphenhydramine; Drug: Ondansetron
- Arm 2, Epley Maneuver (Experimental): Patients will receive vestibular rehabilitation (the Epley Maneuver).
  Interventions: Other: Epley Maneuver

INTERVENTIONS:
Drug: Meclizine — medication administration 25mg PO one time
  Other Names: Antivert
  Arms: Arm 1, Conventional Therapy
Other: Epley Maneuver — Patient has vestibular rehabilitation utilizing the Epley Maneuver.
  Other Names: Canalith Repositioning Technique
  Arms: Arm 2, Epley Maneuver
Drug: Lorazepam — Lorazepam 1 - 5mg PO/IV prn
  Other Names: Valium
  Arms: Arm 1, Conventional Therapy
Drug: Diphenhydramine — 25 - 50mg PO/IV once prn
  Other Names: Benedryl
  Arms: Arm 1, Conventional Therapy
Drug: Ondansetron — Ondansetron 4 - 8 mg PO/IV prn
  Other Names: Zofran
  Arms: Arm 1, Conventional Therapy

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is a common complaint of emergency department patients. The importance of early diagnosis and treatment can lead to a much improved quality of life for patients afflicted by this ailment. It is the purpose of this study to evaluate and examine two methods of treatment. Patients will be randomized to receive the more common conventional medication therapy versus the canalith repositioning technique. All patients enrolled into this study are emergency department patients who have been diagnosed with BPPV via a positive Dix-Hallpike Maneuver. The hypothesis of this study is that vestibular rehabilitation will allow for resolution of symptoms without the use of conventional medication therapy in the acute management of BPPV in the emergency department patient.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV) is the most common peripheral vestibular disorder, accounting for 20% of all vertigo cases. It was first described by Barany in 1921, and later described in more detail by Dix and Hallpike in 1952. Common practice by ED physicians is to rule out serious medical causes for their symptoms. It is presently common for ED physicians to treat these patients mainly with benzodiazepines, antihistamines, and anticholinergic medications, especially if the history and physical is consistent with BPPV. This method of treatment has had questionable success. Several reviews of the management of vertigo have shown that no medication in current use has well established curative or prophylactic value or is suitable for long-term treatment.

The purpose of this study is to compare the efficacy of vestibular rehabilitation vs. conventional therapy in ED patients who present with vertigo. The objectives to be determined in this study are as follows:

Objectives:

1. To evaluate the improvement of vertigo in patients diagnosed with BPPV in the ED.
2. To evaluate disposition time for those patients receiving vestibular rehabilitation in the ED compared to those patients who receive conventional therapy.
3. To demonstrate the long-term improvement of symptomatology utilizing vestibular rehabilitation versus conventional therapy.
4. Compare patient satisfaction between those patients who receive standard care vs. those who receive vestibular rehabilitation.

Inclusion Criteria:

1. Subject is a male or female >18 years of age.
2. Subject has presented to the Emergency Department Monday through Friday during the hours of 8 AM to 4:30 PM or possibly extended into the evening and weekend hours if research or physical therapy staff is available, and is diagnosed with BPPV.
3. Subject has positive findings of vertigo and nystagmus when the Dix-Hallpike maneuver is performed during physical examination. A Dix-Hallpike maneuver will be considered positive when the patient experiences nystagmus but resolves or fatigues in less than 60 seconds
4. Informed consent can be obtained for participation in this study.

Exclusion Criteria:

1. Subject has taken any antihistamines or anticholinergics within the past 12 hours.
2. Subjects who are unable to ambulate.
3. Subjects with severe cervical spine disease or known cerebral vascular disease.
4. Any positive findings during the neurological exam during physical examination.
5. Subjects who have negative finding of vertigo and nystagmus when the Dix- Hallpike maneuver is performed by the Physical Therapist or research staff even if the subject had a positive finding of vertigo and nystagmus when the Dix-Hallpike maneuver was performed by the physician or resident.
6. Subjects with a known history of Meniere's Disease.
7. Any cardiac complaints during physical examination or subject has experienced a positive loss of consciousness.
8. Subject has been previously enrolled in this study.
9. Subjects with mental conditions that render them unable to understand the nature,
10. Subjects who are unlikely to comply with the study such as subjects with uncooperative attitude, unlikely to complete follow-up visits, or unlikely to complete the study.
11. Any other condition which would confound or interfere with evaluation or prevent compliance with the study protocol.

Statistical Considerations/Data Analysis:

Statistical analysis will be completed under consult with Health Studies Research. Inter-Rater Reliability analysis will be completed by the physical therapists and nurse researchers prior to the study using video analysis of nystagmus and post-test of technique by a physical therapist certified in vestibular rehabilitation. After enrollment of these subjects a data peak power analysis will be conducted to calculate exact sample size needed to complete this study. This will also give us an indication of the length of time needed to conduct this study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female >18 years of age.
2. Subject has presented to the Emergency Department Monday through Friday during the hours of 8 AM to 4:30 PM or possibly extended into the evening and weekend hours if research or physical therapy staff is available, and is diagnosed with BPPV.
3. Subject has positive findings of vertigo and nystagmus when the Dix-Hallpike maneuver is performed during physical examination. A Dix-Hallpike maneuver will be considered positive when the patient experiences nystagmus but resolves or fatigues in less than 60 seconds
4. Informed consent can be obtained for participation in this study.

Exclusion Criteria:

1. Subject has taken any antihistamines or anticholinergics within the past 12 hours.
2. Subjects who are unable to ambulate.
3. Subjects with severe cervical spine disease or known cerebral vascular disease.
4. Any positive findings during the neurological exam during physical examination.
5. Subjects who have negative finding of vertigo and nystagmus when the Dix- Hallpike maneuver is performed by the Physical Therapist or research staff even if the subject had a positive finding of vertigo and nystagmus when the Dix-Hallpike maneuver was performed by the physician or resident.
6. Subjects with a known history of Meniere's Disease.
7. Any cardiac complaints during physical examination or subject has experienced a positive loss of consciousness.
8. Subject has been previously enrolled in this study.
9. Subjects with mental conditions that render them unable to understand the nature,
10. Subjects who are unlikely to comply with the study such as subjects with uncooperative attitude, unlikely to complete follow-up visits, or unlikely to complete the study.
11. Any other condition which would confound or interfere with evaluation or prevent compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-11; Primary Completion 2010-12 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Burmeister, DO, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD, just publish the study's results.

REFERENCES:
- [Result] Sacco RR, Burmeister DB, Rupp VA, Greenberg MR. Management of benign paroxysmal positional vertigo: a randomized controlled trial. J Emerg Med. 2014 Apr;46(4):575-81. doi: 10.1016/j.jemermed.2013.08.116. Epub 2014 Jan 22. PMID 24462034

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1, Conventional Therapy | Arm 2, Epley Maneuver
Started | 11 | 15
Completed | 11 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: To be included in the study, patients had to be at least 18 years of age, presenting to the ED weekdays during business hours, and have a positive DH test.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Conventional Therapy | Arm 2, Epley Maneuver | Total
Number analyzed (Participants) | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12.6) | 64 (11.2) | 61.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 8 | 5 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Likert Scale for Satisfaction
Description: The Likert Scale measured patient satisfaction on a 0-10 score range (0 = Least Satisfied; 10 = Most Satisfied).
Time Frame: 0 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1, Conventional Therapy | Arm 2, Epley Maneuver
Number analyzed (Participants) | 11 | 15
units on a scale | 9 (1.5) | 9 (1.0)

ADVERSE EVENTS:
Arm/Group | Arm 1, Conventional Therapy | Arm 2, Epley Maneuver
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes